CLINICAL TRIAL: NCT02503280
Title: A Phase I/II, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Transendocardial Injection of Autologous Human Cells (Mesenchymal or the Combination of MSC and Cardiac Stem Cells) in Patients With Chronic Ischemic Left Ventricular Dysfunction and Heart Failure Secondary to Myocardial Infarction.
Brief Title: The Transendocardial Autologous Cells (hMSC) or (hMSC) and (hCSC) in Ischemic Heart Failure Trial.
Acronym: TAC-HFT-II
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has never enrolled any subjects
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, ISCI Director, Chief Science Officer, Senior Assoc. Dean, Louis Lemberg Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20120203
Record Dates: First submitted 2015-05-04; First posted 2015-07-20 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Ischemic Left Ventricular Dysfunction; Myocardial Infarction
Keywords: Cardiovascular; Secondary
MeSH Terms: conditions — Myocardial Infarction; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - Autologous hMSCs (Experimental): Autologous hMSCs: 40 million cells/ml delivered in 0.5 ml injection volumes times 10 injections for a total of 2 x 10^8 (200 million) hMSCs. The Biosense Webster MyoStar NOGA Injection Catheter System will be used in the delivery of the study drug.
  Interventions: Drug: Autologous hMSCs; Device: Biosense Webster MyoStar NOGA Injection Catheter System
- Group B - Autologous Human C-Kit CSCs II (Experimental): Autologous hMSCs PLUS autologous C-Kit hCSCs: Mixture of 39.8 million hMSCs and 0.2 million C-Kit hCSCs/ml delivered in 0.5 ml injection volumes times 10 injections for a total of 1.99 x 10^8 (199 million) hMSCs and 1 million C-Kit hCSCs.The Biosense Webster MyoStar NOGA Injection Catheter System will be used in the delivery of the study drug.
  Interventions: Drug: Autologous Human C-Kit CSCs II; Device: Biosense Webster MyoStar NOGA Injection Catheter System
- Placebo (Placebo Comparator): Placebo (ten 0.5 ml injections of phosphate-buffered saline [PBS] and 1% human serum albumin [HSA]).The Biosense Webster MyoStar NOGA Injection Catheter System will be used in the delivery of the study drug.
  Interventions: Drug: Placebo; Device: Biosense Webster MyoStar NOGA Injection Catheter System

INTERVENTIONS:
Drug: Autologous hMSCs — Autologous hMSCs: 40 million cells/ml delivered in 0.5 ml injection volumes times 10 injections for a total of 2 x 10^8 (200 million) hMSCs.
  Other Names: Autologous Human Mesenchymal Stem Cells (hMSCs)
  Arms: Group A - Autologous hMSCs
Drug: Autologous Human C-Kit CSCs II — Autologous hMSCs PLUS autologous C-Kit hCSCs: Mixture of 39.8 million hMSCs and 0.2 million C-Kit hCSCs/ml delivered in 0.5 ml injection volumes times 10 injections for a total of 1.99 x 10^8 (199 million) hMSCs and 1 million C-Kit hCSCs.
  Other Names: Autologous Human C-Kit Cardiac Stem Cells (CSCs) II
  Arms: Group B - Autologous Human C-Kit CSCs II
Drug: Placebo — Placebo (ten 0.5 ml injections of phosphate-buffered saline [PBS] and 1% human serum albumin [HSA]).
  Arms: Placebo
Device: Biosense Webster MyoStar NOGA Injection Catheter System — Biosense Webster MyoStar NOGA Injection Catheter System will be used to administer the study drug
  Other Names: NOGA

SUMMARY:
Before initiating the full randomized study, a Pilot Safety Phase will be performed. In this phase the composition of cells administered via the Biosense Webster MyoStar NOGA Injection Catheter System will be tested. The randomized portion of the study will be conducted after a full review of the safety data from the pilot Phase by the Data safety monitoring board.

Following the Pilot Phase of five (5) Fifty (50) patients scheduled to undergo cardiac catheterization and meeting all inclusion/exclusion criteria will be evaluated at baseline.

Patients will be randomized in a 2:2:1 ratio to one of three Treatment Strategies.

DETAILED DESCRIPTION:
A Phase I/II, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Transendocardial Injection of Autologous Human Cells (Mesenchymal or the combination of MSC and Cardiac Stem Cells) in Patients With Chronic Ischemic Left Ventricular Dysfunction and Heart Failure Secondary to Myocardial Infarction.

A total of 55 subjects participating, with 5 in the pilot phase and 50 in the randomized phase.

Patients with chronic ischemic left ventricular dysfunction and heart failure secondary to MI scheduled to undergo cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* In order to participate in this study, a patient MUST:

  1. Be ≥ 21 and < 90 years of age.
  2. Provide written informed consent.
  3. Have a diagnosis of chronic ischemic left ventricular dysfunction secondary to myocardial infarction (MI) as defined by the following: Screening MRI must show an area of akinesis, dyskinesis, or severe hypokinesis associated with evidence of myocardial scarring based on delayed hyperenhancement following gadolinium infusion.
  4. Been treated with appropriate maximal medical therapy for heart failure or post-infarction left ventricular dysfunction. For beta-blockade, the patient must have been on a stable dose of a clinically appropriate beta-blocker for 3 months. For angiotensin-converting enzyme inhibition, the patient must have been on a stable dose of a clinically appropriate agent for 1 month.
  5. Be a candidate for cardiac catheterization.
  6. Have an ejection fraction ≤ 50% by gated blood pool scan, two-dimensional echocardiogram, cardiac MRI, or left ventriculogram within the prior six months and not in the setting of a recent ischemic event.

Exclusion Criteria:

* In order to participate in this study, a patient MUST NOT:

  1. Have a baseline glomerular filtration rate < 50 ml/min1.73m2.
  2. Have a known, serious radiographic contrast allergy.
  3. Have a mechanical aortic valve or heart constrictive device.
  4. Have a documented presence of aortic stenosis (aortic stenosis graded as ≥ +2 equivalent to an orifice area of 1.5cm2 or less).
  5. Have a documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥+2).
  6. Require coronary artery revascularization. Patients who require or undergo revascularization procedures should undergo these procedures a minimum of 3 months in advance of treatment within this study. In addition, patients who develop a need for revascularization following enrollment will be submitted for this therapy without delay.
  7. Evidence of a life-threatening arrhythmia (nonsustained ventricular tachycardia ≥ 20 consecutive beats or complete heart block) or QTc interval > 550 ms on screening ECG.
  8. AICD firing in the past 60 days prior to the procedure.
  9. Have unstable angina within 2 weeks of the planned procedure.
  10. Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
  11. Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the ULN.
  12. Have a coagulopathy = (INR > 1.3) not due to a reversible cause (i.e., Coumadin). Patients on Coumadin will be withdrawn 5 days before the procedure and confirmed to have an INR < 1.3. Patients who cannot be withdrawn from Coumadin will be excluded from enrollment
  13. Have known allergies to penicillin or streptomycin.
  14. Have a contra-indication to performance of an MRI scan.
  15. Be an organ transplant recipient.
  16. Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
  17. Have a non-cardiac condition that limits lifespan to < 1 year.
  18. Have a history of drug or alcohol abuse within the past 24 months.
  19. Be on chronic therapy with immunosuppressant medication, such as corticosteroids or TNFα antagonists.
  20. Be serum positive for HIV, hepatitis BsAg or hepatitis C.
  21. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
  22. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of any treatment emergent serious adverse events (TE-SAEs) | One Month post-catheterization
  Incidence (at one month post-catheterization) of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of: death, non-fatal MI, stroke, hospitalization for worsening heart failure, cardiac perforation, pericardial tamponade, sustained ventricular arrhythmias (characterized by ventricular arrhythmias lasting longer than 15 seconds or with hemodynamic compromise), or atrial fibrillation.

SECONDARY OUTCOMES:
Treatment Emergent adverse event rates | At 6 Month and 12 Month visit
  Rate of adverse events occurring ad
Ectopic tissue formation | At 6 Month and 12 Month visit
  Ectopic tissue formation (as identified from MRI scans of the chest, abdomen, & pelvis).
48-hour ambulatory electrocardiogram (ECG) recordings. | At 6 Month and 12 Month visit
  Electrocardiogram (ECG) recordings measured over 48 Hours
Hematology value changes post-catheterization | At 6 Month and 12 Month visit
  Hematology value changes will be observed at the 6 month and 12 month visit post-catheterization.
Urinalysis results changes post-catheterization | At 6 Month and 12 Month visit
  Urinalysis results changes will be observed at the 6 month and 12 month visit post-catheterization.
Clinical chemistry values post-catheterization | At 6 Month and 12 Month visit
  Clinical chemistry value changes will be observed at the 6 month and 12 month visit post-catheterization.
Pulmonary function | At 6 Month and 12 Month visit
  Pulmonary function - forced expiratory volume in 1 second (FEV1) results.
Serial troponin I values | Every 12 hours for the first 48 hours post-cardiac catheterization
  Serial troponin I values (every 12 hours for first 48 hours post-cardiac catheterization).
Creatine kinase-MB (CK-MB) value changes post-catheterization | Every 12 hours for first 48 hours post-cardiac catheterization
  CK-MB values (every 12 hours for first 48 hours post-cardiac catheterization).
Post-cardiac catheterization echocardiogram. | Day 1 Post Echocardiogram
  Echocardiogram performed after cardiac catheterization
Magnetic resonance imaging (MRI) measures of infarct scar size (ISS) | At 6 Month and 12 Month visit
  Document Infarct Scar Size (ISS) via Magnetic Resonance imaging (MRI)
Echocardiographic measures of infarct scar size (ISS) | At 6 Month and 12 Month visit
  Document Infarct Scar Size (ISS) via echocardiographic procedure
Magnetic resonance imaging (MRI) of Left Regional Ventricular Function | At 6 Month and 12 Month visit
  Document Left Regional Ventricular Function via Magnetic Resonance imaging (MRI)
Echocardiographic measures of Left Regional Ventricular Function | At 6 Month and 12 Month visit
  Document Left Regional Ventricular Function via echocardiographic procedure
Magnetic resonance imaging (MRI) of Global Ventricular Function | At 6 Month and 12 Month visit
  Document Global Ventricular Function via Magnetic Resonance imaging (MRI)
Echocardiographic measures of Global Ventricular Function | At 6 Month and 12 Month visit
  Document Global Ventricular Function via echocardiographic procedure
Tissue perfusion measured by MRI. | At 6 Month and 12 Month visit
  Measure Tissue Perfusion via Magnetic Resonance imaging (MRI)
Peak oxygen consumption (Peak VO2) (by treadmill determination). | At 6 Month and 12 Month visit
  Peak VO2 Oxygen Consumption determined by utilizing treadmill
Six-minute walk test. | At 6 Month and 12 Month visit
  Evaluate Functional Capacity via the Six Minute Walk Test
New York Heart Association (NYHA) functional class. | At 6 Month and 12 Month visit
  Evaluate Functional Capacity via New York Heart Association (NYHA) Class Determination
Minnesota Living with Heart Failure (MLHF) questionnaire. | At 6 Month and 12 Month visit
  Evaluate Quality Of Life Changes via Minnesota Living with Heart Failure (MLHF) Questionnaire
Incidence of Major Adverse Cardiac Events (MACE) | At 6 Month and 12 Month visit
  Incidence of Major Adverse Cardiac Events (MACE), defined as the composite incidence of (1) death, (2) hospitalization for worsening HF, or (3) non-fatal recurrent MI.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI / University of Miami Miller School of Medicine
Locations (1):
- ISCI / University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School of Medicine — http://isci.med.miami.edu